CLINICAL TRIAL: NCT05044923
Title: Restoring Hemodynamic Stability Using Targeted Epidural Spinal Stimulation Following Spinal Cord Injury
Acronym: HEMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aaron Phillips (Other)
Responsible Party: Sponsor-Investigator, Aaron Phillips, Assistant Professor, University of Calgary
Organization: University of Calgary (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB21-0027
Record Dates: First submitted 2021-08-27; First posted 2021-09-16 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Spinal Cord Injuries
Keywords: orthostatic hypotension; autonomic dysreflexia; epidural stimulation; blood pressure
MeSH Terms: conditions — Spinal Cord Injuries; Hypotension, Orthostatic; Autonomic Dysreflexia

STUDY DESIGN:
Intervention Model Description: Single-site, single-are, non-blinded, non-randomized, interventional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Targeted Epidural Spinal Stimulation (Experimental): Participants will undergo surgery to implant devices that will be used for Targeted Epidural Spinal Stimulation (TESS).
  Interventions: Device: Targeted Epidural Spinal Stimulation

INTERVENTIONS:
Device: Targeted Epidural Spinal Stimulation — Two lead electrodes (Specify Surescan 5-6-5 Leads, Model 977C190 Medtronic) will be implanted epidurally over the dorsal aspect of the spinal cord through two laminotomies. Two implantable pulse generators (Intellis™ with AdaptiveStim™, Model 97715 Medtronic) will be connected to the lead electrodes and implanted in the upper buttocks of the participant.

SUMMARY:
The purpose of this study is to stimulate the circuits in the spinal cord that are directly responsible for hemodynamic control to restore hemodynamic stability in participants with chronic cervical or high-thoracic spinal cord injury. The ultimate objective of this study is to provide preliminary safety and efficacy measures on the ability of the hemodynamic Targeted Epidural Spinal Stimulation (TESS) to ensure the long-term management of hemodynamic instability and reduce the incidence and severity of orthostatic hypotension and autonomic dysreflexia episodes in individuals with chronic cervical or high-thoracic spinal cord injury. In addition, the long-term safety and efficacy of TESS on cardiovascular health, respiratory function, and quality of life in participants with chronic spinal cord injury will be evaluated.

DETAILED DESCRIPTION:
Clinical management of chronic hemodynamic instability is currently limited to long-acting pressor agents and anti-hypertensives. These drugs have significant limitations as they require roughly one hour to become active and exert prolonged influences on the cardiovascular system. This slow timescale contrasts with the hemodynamic instability experienced by people with spinal cord injury, which occurs most commonly over just a few minutes, and tends to cease abruptly. This study will investigate a new therapy for managing hemodynamic instability in individuals with spinal cord injury: Targeted Epidural Spinal Stimulation (TESS).

Here, the investigators propose to stimulate the circuits in the spinal cord that are directly responsible for hemodynamic control to restore hemodynamic stability in participants with chronic cervical or high-thoracic spinal cord injury. The ultimate objective of this feasibility study is to provide preliminary safety and efficacy measures on the ability of the hemodynamic TESS to ensure the long-term management of hemodynamic instability and reduce the incidence and severity of orthostatic hypotension and autonomic dysreflexia episodes in humans with chronic cervical or high-thoracic spinal cord injury. In addition, the investigators aim to evaluate the long-term safety and efficacy of TESS on cardiovascular health, respiratory function, spasticity, trunk stability, sleep and quality of life in participants with chronic spinal cord injury.

The HEMO Trial will implant 4 participants with chronic (>12 months) spinal cord injury located between C3 and T6 who have confirmed severe orthostatic hypotension and autonomic dysreflexia. Enrolled participants will undergo baseline assessments, after which they will be implanted with the investigational system. Participants will then proceed to one month of an intensive device configuration protocol to configure the TESS settings of their investigational device to regain hemodynamic stability. After the intensive device configuration phase, daily supervised at-home hemodynamic TESS will be conducted for two weeks. Thereafter, and up to 25 weeks post-implant, participants will conduct supported at-home sessions as well as regular laboratory visits during a long-term at-home hemodynamic TESS phase. Finally, participants will undergo additional testing during a configuration of additional TESS programs phase. During this phase TESS configurations for hemodynamic stability, respiratory function, trunk stability and spasticity will be tested. Several clinical evaluations are planned to evaluate participants' hemodynamic and neurological status, cardiovascular functional status, respiratory function, trunk stability, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years old
* Able to undergo the informed consent/assent process
* Radiologically confirmed spinal cord injury
* Spinal cord injury between C3 and T6
* Classified with American Spinal Injury Association Impairment Scale (AIS) A or B Spinal cord injury
* Stable medical, physical and psychological condition as considered by Investigators
* Greater than 1 year since initial injury and at least 6 months from any required spinal instrumentation
* Confirmed orthostatic hypotension and autonomic dysreflexia
* Willing to attend all scheduled appointments

Exclusion Criteria:

* Diseases and conditions that would increase the morbidity and mortality of spinal cord injury surgery
* The inability to withhold antiplatelet/anticoagulation agents perioperatively
* History of myocardial infarction or cerebrovascular event
* Other conditions that would make the subject unable to participate in testing in the judgment of the investigators
* Current and anticipated need for opioid pain medications or pain that would prevent full participation in the trial in the judgement of the investigators
* Current clinical diagnosis of mental illness
* Clinically significant cognitive impairment
* Current substance or alcohol abuse
* Botulinum toxin injections in the previous 6 months
* Presence of significant pressure ulcers
* Recurrent urinary tract infection refractory to antibiotics
* Current pregnancy
* Current breast feeding
* Unhealed spinal fractures
* Presence of indwelling baclofen or insulin pump

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Adverse Events and Serious Adverse Events that are deemed related or possibly related to the study procedure or to the study investigational system, from implant surgery until the end of study | From implant surgery through study completion, an average of 7 months
  Investigate the preliminary safety of hemodynamic targeted epidural spinal stimulation (TESS) to modulate pressor responses and manage blood pressure instability in participants with chronic SCI located between C3 and T6 and who suffer from severe orthostatic hypotension.

SECONDARY OUTCOMES:
Orthostatic head-up tilt test | At baseline and during the testing phase, an average of 9 months
  Beat-by-beat blood pressure is recorded as participants are passively tilted from a supine position to an upright position using a motorized table.
Daily stimulation log | From implant surgery through study completion, an average of 7 months
  Participants will self-report the use of Targeted Epidural Spinal Stimulation (TESS).
Echocardiogram (Ejection Fraction) | At baseline and during the testing phase, an average of 9 months
  Ultrasound will be used to assess cardiac structure and function. Ejection fraction will be recorded.
Echocardiogram (Strain) | At baseline and during the testing phase, an average of 9 months
  Ultrasound will be used to assess cardiac structure and function. Global longitudinal strain will be recorded.
Vascular ultrasound | At baseline and during the testing phase, an average of 9 months
  Flow-mediated dilation assessments will be performed using ultrasound to assess vascular structure and function.
Autonomic Dysfunction Following Spinal Cord Injury (ADFSCI) Questionnaire | At baseline and during the testing phase, an average of 9 months
  The ADFSCI is a 24-item self-report questionnaire. The questionnaire consists of demographics, medications, frequency/severity of symptoms during AD and hypotensive events. Higher scores indicate greater severity and frequency of AD episodes.
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) | At baseline and during the testing phase, an average of 9 months
  Clinical examination used to assess the motor and sensory impairment and severity of a spinal cord injury.
Respiratory function evaluation (Volume) | At baseline and during the testing phase, an average of 9 months
  Respiratory function will be assessed using a spirometer while the participant performs a systematic set of breathing tasks. Volume will be recorded.
Respiratory function evaluation (Flow) | At baseline and during the testing phase, an average of 9 months
  Respiratory function will be assessed using a spirometer while the participant performs a systematic set of breathing tasks. Flow will be recorded.
Quality of life questionnaire (WHOQOL-BREF) | At baseline and during the testing phase, an average of 9 months
  The WHOQOL-BREF is a 26-item self-report questionnaire. The questionnaire covers physical and psychological health, social relationships, and environment. Higher scores indicate higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Phillips, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Squair JW, Gautier M, Mahe L, Soriano JE, Rowald A, Bichat A, Cho N, Anderson MA, James ND, Gandar J, Incognito AV, Schiavone G, Sarafis ZK, Laskaratos A, Bartholdi K, Demesmaeker R, Komi S, Moerman C, Vaseghi B, Scott B, Rosentreter R, Kathe C, Ravier J, McCracken L, Kang X, Vachicouras N, Fallegger F, Jelescu I, Cheng Y, Li Q, Buschman R, Buse N, Denison T, Dukelow S, Charbonneau R, Rigby I, Boyd SK, Millar PJ, Moraud EM, Capogrosso M, Wagner FB, Barraud Q, Bezard E, Lacour SP, Bloch J, Courtine G, Phillips AA. Neuroprosthetic baroreflex controls haemodynamics after spinal cord injury. Nature. 2021 Feb;590(7845):308-314. doi: 10.1038/s41586-020-03180-w. Epub 2021 Jan 27. PMID 33505019
- [Background] Anderson KD. Targeting recovery: priorities of the spinal cord-injured population. J Neurotrauma. 2004 Oct;21(10):1371-83. doi: 10.1089/neu.2004.21.1371. PMID 15672628
- [Background] Cragg JJ, Noonan VK, Krassioukov A, Borisoff J. Cardiovascular disease and spinal cord injury: results from a national population health survey. Neurology. 2013 Aug 20;81(8):723-8. doi: 10.1212/WNL.0b013e3182a1aa68. Epub 2013 Jul 24. PMID 23884034
- [Background] Illman A, Stiller K, Williams M. The prevalence of orthostatic hypotension during physiotherapy treatment in patients with an acute spinal cord injury. Spinal Cord. 2000 Dec;38(12):741-7. doi: 10.1038/sj.sc.3101089. PMID 11175374
- [Background] Phillips AA, Krassioukov AV. Contemporary Cardiovascular Concerns after Spinal Cord Injury: Mechanisms, Maladaptations, and Management. J Neurotrauma. 2015 Dec 15;32(24):1927-42. doi: 10.1089/neu.2015.3903. Epub 2015 Sep 1. PMID 25962761
- [Background] Phillips AA, Krassioukov AV, Ainslie PN, Warburton DE. Perturbed and spontaneous regional cerebral blood flow responses to changes in blood pressure after high-level spinal cord injury: the effect of midodrine. J Appl Physiol (1985). 2014 Mar 15;116(6):645-53. doi: 10.1152/japplphysiol.01090.2013. Epub 2014 Jan 16. PMID 24436297
- [Background] Phillips AA, Warburton DE, Ainslie PN, Krassioukov AV. Regional neurovascular coupling and cognitive performance in those with low blood pressure secondary to high-level spinal cord injury: improved by alpha-1 agonist midodrine hydrochloride. J Cereb Blood Flow Metab. 2014 May;34(5):794-801. doi: 10.1038/jcbfm.2014.3. Epub 2014 Jan 29. PMID 24473484
- [Background] Phillips AA, Elliott SL, Zheng MM, Krassioukov AV. Selective alpha adrenergic antagonist reduces severity of transient hypertension during sexual stimulation after spinal cord injury. J Neurotrauma. 2015 Mar 15;32(6):392-6. doi: 10.1089/neu.2014.3590. Epub 2014 Dec 5. PMID 25093677
- [Background] Krassioukov A, Eng JJ, Warburton DE, Teasell R; Spinal Cord Injury Rehabilitation Evidence Research Team. A systematic review of the management of orthostatic hypotension after spinal cord injury. Arch Phys Med Rehabil. 2009 May;90(5):876-85. doi: 10.1016/j.apmr.2009.01.009. PMID 19406310
- [Background] Squair JW, Phillips AA, Harmon M, Krassioukov AV. Emergency management of autonomic dysreflexia with neurologic complications. CMAJ. 2016 Oct 18;188(15):1100-1103. doi: 10.1503/cmaj.151311. Epub 2016 May 24. No abstract available. PMID 27221275
- [Background] Phillips AA, Krassioukov AV, Ainslie PN, Warburton DE. Baroreflex function after spinal cord injury. J Neurotrauma. 2012 Oct 10;29(15):2431-45. doi: 10.1089/neu.2012.2507. Epub 2012 Sep 20. PMID 22897489
- [Background] Courtine G, Gerasimenko Y, van den Brand R, Yew A, Musienko P, Zhong H, Song B, Ao Y, Ichiyama RM, Lavrov I, Roy RR, Sofroniew MV, Edgerton VR. Transformation of nonfunctional spinal circuits into functional states after the loss of brain input. Nat Neurosci. 2009 Oct;12(10):1333-42. doi: 10.1038/nn.2401. Epub 2009 Sep 20. PMID 19767747
- [Background] Wagner FB, Mignardot JB, Le Goff-Mignardot CG, Demesmaeker R, Komi S, Capogrosso M, Rowald A, Seanez I, Caban M, Pirondini E, Vat M, McCracken LA, Heimgartner R, Fodor I, Watrin A, Seguin P, Paoles E, Van Den Keybus K, Eberle G, Schurch B, Pralong E, Becce F, Prior J, Buse N, Buschman R, Neufeld E, Kuster N, Carda S, von Zitzewitz J, Delattre V, Denison T, Lambert H, Minassian K, Bloch J, Courtine G. Targeted neurotechnology restores walking in humans with spinal cord injury. Nature. 2018 Nov;563(7729):65-71. doi: 10.1038/s41586-018-0649-2. Epub 2018 Oct 31. PMID 30382197